CLINICAL TRIAL: NCT01286844
Title: An Open Label, Dose Escalation Study to Examine the Pharmacokinetics, Pharmacodynamics and Safety and Tolerability of Single and Repeat Oral Doses of GSK2190915 in Children Aged From 1 to 11 Years With Asthma
Brief Title: GSK2190915 Pediatric Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112361
Record Dates: First submitted 2010-10-07; First posted 2011-01-31 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects ≥4 and< 12 years. First 6 subjects included, ≥8 and< 12 yrs and weigh ≥21kg, receive 1 SD (10mg) and an 8 day RD period (100mg). Remaining subjects in cohort: Subjects < 21kg receive 2 SD periods (10mg and 50mg), Subjects > 21kg receive 2 SD periods (10mg and 50mg) and an 8 day RD (100mg)
  Interventions: Drug: GSK2190915A 10mg; Drug: GSK2190915A 50mg; Drug: GSK2190915A 100mg
- Cohort 2 (Experimental): Subjects ≥1 and< 4 years, receive 2 SD (5mg and 25mg)
  Interventions: Drug: GSK2190915A 5mg; Drug: GSK2190915A 25mg

INTERVENTIONS:
Drug: GSK2190915A 5mg — Oral powder for dispersion in water
  Arms: Cohort 2
Drug: GSK2190915A 10mg — Oral powder for dispersion in water
  Arms: Cohort 1
Drug: GSK2190915A 25mg — Oral powder for dispersion in water
  Arms: Cohort 2
Drug: GSK2190915A 50mg — Oral powder for dispersion in water
  Arms: Cohort 1
Drug: GSK2190915A 100mg — Oral powder for dispersion in water
  Arms: Cohort 1

SUMMARY:
GSK2190915 is under development as an oral controller for the treatment of adult and pediatric asthma. This study is an open label, single and repeat dose escalation study, in children with asthma. It will investigate the pharmacokinetics of GSK2190915 in children, aged from 1 to 12 years old inclusive, to determine how the dosage regimen for GSK2190915 in a pediatric population should be adjusted to achieve approximately the same level of systemic exposure that is safe and effective in adults.

DETAILED DESCRIPTION:
Subjects will be recruited into 2 cohorts, Cohort 1 with children from 4 years of age to less than 12 years of age and cohort 2 with children from 1 year of age to less than 4 years of age. Cohort 1 is further subdivided, dependent on a subject's weight, which enables different dosing regimens and pharmacokinetic sampling within the cohort. There are 3 scheduled Pharmacokinetic and Safety Review meetings, which enable dose adjustment and dosing in the younger subjects through the study.

Blood and urine are collected for pharmacokinetic and pharmacodynamic analysis. Safety will be assessed by measurement of heart rate, blood pressure, ECG, safety laboratory data and review of adverse events. Subjects will also perform PEF and Spirometry if assessed as capable by the study investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male and pre-menarchial female subjects aged 1to <12 years at screening are eligible for this study.
* Investigator diagnosed history of asthma.
* Subject weight a minimum of 11kg and above the 10th percentile for their age.
* Patients must be controlled on any existing asthma treatment or currently stable off treatment, at screening.
* Apart from asthma, eczema and rhinitis, subjects should be healthy and suffer from no other significant medical conditions.
* Subjects and parents/guardians must be able to understand and comply with protocol requirements, instructions and protocol-stated restrictions. Parents/guardians must have the ability to read and write.

A signed and dated informed consent from at least one parent/guardian, and, for subjects ≥ 7 years old an accompanying informed assent from the subject prior to admission to the study.

- AST and ALT < 2xULN.

Exclusion Criteria:

* Subjects who have changed their asthma medication, dose or regime within 4 weeks of screening
* Administration of anti -leukotriene therapies for 14 days before screening and during the study.
* Any medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Any clinically relevant abnormality identified on the screening medical assessment.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of screening and led to a change in asthma management.
* Administration of any vaccinations within 2 weeks of screening or during the study
* Parent/guardian has history of psychiatric disease, intellectual deficiency, substance abuse, or other condition which will limit the validity of consent to participate in this study.
* Any adverse reaction including immediate or delayed hypersensitivity to any component of study drug
* A subject will not be eligible for this study if he/she is an immediate family member of the participating Investigator, sub-Investigator, study coordinator, or employee of the participating Investigator.
* Children who are wards of the state or government.
* The subject has a screening QTc value of >450msec, PR interval outside the range 120 to 220msec or an ECG that is not suitable for QT measurements.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Derived plasma pharmacokinetic parameters | 24 hours

SECONDARY OUTCOMES:
Leukotriene biomarkers | 24 hours
Vital Signs | 24 hours
ECG | 24 hours
Adverse Event Monoitoring | Up to 90 days
Clinical Labs | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline